CLINICAL TRIAL: NCT06194617
Title: The Exploratory Study on Clinical Rational Use of Rivaroxaban Dosing in Elderly Chinese Population
Brief Title: Rivaroxaban in Elderly Chinese Venous Thromboembolism Patients
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-Rivaroxaban in Elderly
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism; Anticoagulant-induced Bleeding
Keywords: Pulmonary Embolism; Venous Thromboembolism; Direct Oral Anticoagulants
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood and Urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with pulmonary embolism and using direct oral anticoagulants: Patients with pulmonary embolism and using direct oral anticoagulants
  Interventions: Drug: Direct oral anticoagulant

INTERVENTIONS:
Drug: Direct oral anticoagulant — Patients take DOACs according to their condition, with the dosage determined by the clinical physician.

SUMMARY:
There's no unified recommendation in clinical practice regarding adjusting dosages for different patient types, especially when adverse events occur. While rivaroxaban typically doesn't require coagulation monitoring, in elderly patients, particularly those with multiple medications, finding appropriate lab indicators becomes crucial to gauge its anticoagulant effect. This aids in evaluating precise rivaroxaban dosing for the elderly, balancing bleeding risks and recurrence. Clinical pharmacological studies suggest that drug pharmacokinetics and pharmacodynamics in different populations can guide dosage optimization. Hence, this study aims to provide a basis for optimizing dosing regimens in high-risk elderly patients in China by exploring pharmacokinetic and pharmacodynamic indicators in clinical practice.

DETAILED DESCRIPTION:
Comparison between the traditional anticoagulant warfarin and novel oral anticoagulants reveals the predictable pharmacokinetic and pharmacodynamic characteristics of the latter, with minimal influence from food and other medications, often eliminating the need for routine coagulation monitoring. As a representative of these novel oral anticoagulants, the Xa factor inhibitor rivaroxaban is widely used in the anticoagulant therapy of pulmonary embolism patients. Common adverse events associated with rivaroxaban include severe blood clots (such as pulmonary embolism) and bleeding events. This medication undergoes hepatic and renal dual-mode metabolism, with drug concentrations being influenced by both liver and kidney function. Studies indicate that in patients with impaired kidney function, using the recommended dose can lead to overdosing and increased risk of bleeding. Guidelines suggest that patients with mild renal impairment (creatinine clearance 50-80 mL/min) or moderate renal impairment (creatinine clearance 30-49 mL/min) do not require adjustment of rivaroxaban doses. For patients with severe renal impairment (creatinine clearance 15-29 mL/min), limited clinical data suggests significantly elevated blood drug concentrations with rivaroxaban, indicating its avoidance. For patients with impaired liver function: rivaroxaban is contraindicated in patients with coagulation abnormalities and clinically relevant bleeding risks, including those with Child-Pugh B and C stage cirrhosis. CYP3A4 and P-gp inhibitors elevate rivaroxaban blood concentrations, particularly evident in cases of renal impairment.

Elderly patients, characterized by declining renal function with age, multiple comorbidities, and polypharmacy, exhibit numerous uncertainties, often experiencing either over-anticoagulation or inadequate anticoagulation. Phase I clinical studies of rivaroxaban in healthy elderly individuals confirmed significant increases in pharmacodynamic parameters (Xa factor inhibition rate, PT) compared to younger individuals. The AUC (area under the curve) of Xa factor inhibition rate in the elderly was 41% higher than in younger individuals. This study attributed the results to declining renal function in the elderly. Population pharmacokinetic studies also confirm that after the age of 65, the complete clearance rate of rivaroxaban decreases annually by 1.05-1.5%.

Therefore, there's no unified recommendation in clinical practice regarding the necessity of adjusting corresponding dosing regimens in different patient types, especially when adverse events occur. While rivaroxaban typically does not require coagulation monitoring in most cases, in elderly patients, particularly those on multiple medications, there is a clinical need to identify suitable laboratory monitoring indicators to measure its anticoagulant efficacy, further assessing the optimal dosage for the elderly population to balance bleeding and recurrence risks. Clinical pharmacological studies indicate that the pharmacokinetic and pharmacodynamic characteristics of drugs in different populations can provide a basis for optimizing dosing regimens. Thus, this study aims to provide a basis for optimizing dosing regimens in the clinical practice of elderly high-risk patients in China through an exploration of the pharmacokinetic and pharmacodynamic indicators.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adult patients with objectively diagnosed acute symptomatic pulmonary embolism (with or without concurrent deep vein thrombosis) by imaging, who have completed acute anticoagulation and entered the anticoagulation maintenance phase; (2) Life expectancy greater than 3 months; (3) Meeting the indications for Xa factor inhibitor use; (4) Willingness to participate in this study, sign the informed consent form, and adhere to regular follow-ups.

Exclusion Criteria:

* (1) Moderate or severe hepatic impairment (Child-Pugh Class B or C); (2) Severe renal impairment (CrCl < 15ml/min); (3) Pregnant or breastfeeding women; (4) Spontaneous bleeding tendencies, such as coagulation disorders or low platelet count (PLT < 20×10^9/L); (5) Contraindications to other Xa factor inhibitors' usage; (6) Patients diagnosed with hereditary thrombophilia and antiphospholipid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with objectively diagnosed acute symptomatic pulmonary embolism (with or without concurrent deep vein thrombosis) by imaging, who have completed acute anticoagulation and entered the anticoagulation maintenance phase。
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Symptomatic recurrence of VTE. | through study completion, an average of 1 year
  Recurrent VTE.
Fatal or non-fatal PTE. | through study completion, an average of 1 year
  Recurrent VTE.
Major bleeding (MB) and clinically relevant non-major bleeding (CRNMB) events as defined by the International Society on Thrombosis and Haemostasis (ISTH). | through study completion, an average of 1 year
  Bleeding Events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China